CLINICAL TRIAL: NCT00069511
Title: 12 Week Study of Anti-Viral Effect of Oral UT-231B in Non-cirrhotic Hepatitis C Patients who have Failed Interferon-based Therapy.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: United Therapeutics (Industry)
Organization: Unither Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UT-231B-02:01
Record Dates: First submitted 2003-09-29; First posted 2003-09-30 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-06

CONDITIONS: Hepatitis C
Keywords: Hepatitis C
MeSH Terms: conditions — Hepatitis C

INTERVENTIONS:
Drug: UT-231B

SUMMARY:
This is a multi-center study. Neither the study subjects nor the physicians will know what treatment an individual subject is receiving. Subjects will be randomly assigned (like flipping a coin) to one of five treatment groups. The treatment groups include four different dosing groups of active study drug and one group of subjects who will receive placebo. A 12 week follow up period occurs after the 12 weeks of dosing. The study endpoint is a reduction in Hepatitis C viral load.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be adults,
* have a positive Hepatitis C antibody test,
* and be genotype 1, with a minimum of 100,000 IU of Hepatitis C virus by nucleic acid testing, be non-cirrhotic with a Metavir score of F0-3 (or equivalent) on liver biopsy, and have failed previous therapy with Interferon or Peg Interferon monotherapy, Interferon plus ribavirin, or Peg Interferon and ribavirin.

Exclusion Criteria:

* Diabetics are excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72
Dates: Start 2003-07; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Overall Officials: Katrina L Swartz, PA-C, MHS, Study Director — United Therapeutics
Locations (6):
- United States (6):
  - Shands Hospital at the University of Florida, Gainesville, Florida
  - Tulane Univ. Health Sciences Center, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - UNC Hospital, Chapel Hill, North Carolina
  - Memphis Gastroenterology Group, Memphis, Tennessee
  - VCU/MCV, Richmond, Virginia

REFERENCES:
- [Background] Rosen HR, Martin P. Hepatitis B and C in the liver transplant recipient. Semin Liver Dis. 2000;20(4):465-80. doi: 10.1055/s-2000-13156. PMID 11200416
- [Background] Durantel D, Branza-Nichita N, Carrouee-Durantel S, Butters TD, Dwek RA, Zitzmann N. Study of the mechanism of antiviral action of iminosugar derivatives against bovine viral diarrhea virus. J Virol. 2001 Oct;75(19):8987-98. doi: 10.1128/JVI.75.19.8987-8998.2001. PMID 11533162
- [Background] Pavlovic D, Neville DC, Argaud O, Blumberg B, Dwek RA, Fischer WB, Zitzmann N. The hepatitis C virus p7 protein forms an ion channel that is inhibited by long-alkyl-chain iminosugar derivatives. Proc Natl Acad Sci U S A. 2003 May 13;100(10):6104-8. doi: 10.1073/pnas.1031527100. Epub 2003 Apr 28. PMID 12719519
- [Background] Chylack LT Jr, Wolfe JK, Singer DM, Leske MC, Bullimore MA, Bailey IL, Friend J, McCarthy D, Wu SY. The Lens Opacities Classification System III. The Longitudinal Study of Cataract Study Group. Arch Ophthalmol. 1993 Jun;111(6):831-6. doi: 10.1001/archopht.1993.01090060119035. PMID 8512486
- [Background] Karbassi M, Khu PM, Singer DM, Chylack LT Jr. Evaluation of lens opacities classification system III applied at the slitlamp. Optom Vis Sci. 1993 Nov;70(11):923-8. doi: 10.1097/00006324-199311000-00009. PMID 8302528
- [Background] Ross RS, Viazov S, Sarr S, Hoffmann S, Kramer A, Roggendorf M. Quantitation of hepatitis C virus RNA by third generation branched DNA-based signal amplification assay. J Virol Methods. 2002 Mar;101(1-2):159-68. doi: 10.1016/s0166-0934(01)00433-5. PMID 11849694
- [Background] Lauer GM, Walker BD. Hepatitis C virus infection. N Engl J Med. 2001 Jul 5;345(1):41-52. doi: 10.1056/NEJM200107053450107. No abstract available. PMID 11439948
- [Background] Alter MJ, Kruszon-Moran D, Nainan OV, McQuillan GM, Gao F, Moyer LA, Kaslow RA, Margolis HS. The prevalence of hepatitis C virus infection in the United States, 1988 through 1994. N Engl J Med. 1999 Aug 19;341(8):556-62. doi: 10.1056/NEJM199908193410802. PMID 10451460
- [Background] France MR. Hepatitis C Therapy 2002. Advance for Physician Assistants 2002;10:60-75.
- [Background] Schiff ER, McHutchison JG, Jacobson IM, Lindsay KL, Bacon BR, Maddrey WC. Confronting the Growing Threat of Hepatitis C: a New Call to Action. The Treatment Reporter: Gastroenterology. Secaucus, NJ: Projects in Knowledge Inc.; 2000.
- [Background] Zeuzem S, Feinman SV, Rasenack J, Heathcote EJ, Lai MY, Gane E, O'Grady J, Reichen J, Diago M, Lin A, Hoffman J, Brunda MJ. Peginterferon alfa-2a in patients with chronic hepatitis C. N Engl J Med. 2000 Dec 7;343(23):1666-72. doi: 10.1056/NEJM200012073432301. PMID 11106715
- [Background] Manns MP, McHutchison JG, Gordon SC, Rustgi VK, Shiffman M, Reindollar R, Goodman ZD, Koury K, Ling M, Albrecht JK. Peginterferon alfa-2b plus ribavirin compared with interferon alfa-2b plus ribavirin for initial treatment of chronic hepatitis C: a randomised trial. Lancet. 2001 Sep 22;358(9286):958-65. doi: 10.1016/s0140-6736(01)06102-5. PMID 11583749
- [Background] Fried MW, Shiffman ML, Reddy KR, Smith C, Marinos G, Goncales FL Jr, Haussinger D, Diago M, Carosi G, Dhumeaux D, Craxi A, Lin A, Hoffman J, Yu J. Peginterferon alfa-2a plus ribavirin for chronic hepatitis C virus infection. N Engl J Med. 2002 Sep 26;347(13):975-82. doi: 10.1056/NEJMoa020047. PMID 12324553
- [Background] McHutchison JG. Hepatitis C advances in antiviral therapy: what is accepted treatment now? J Gastroenterol Hepatol. 2002 Apr;17(4):431-41. doi: 10.1046/j.1440-1746.2002.02777.x. PMID 11982724
- See also: trial listing service with patient screener and call center — http://www.veritasmedicine.com